CLINICAL TRIAL: NCT00760981
Title: A Pilot Study of Imatinib Mesylate in Steroid Refractory Chronic Graft Versus Host Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: David Miklos (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, David Miklos, Assistant Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-14821; 14821 (Other: Stanford University Alternate IRB Approval Number); BMT195 (Other: OnCore Number)
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Graft vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Imatinib (Experimental): 200 mg orally daily and 400 mg orally daily for 4 weeks.
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — The single cohort for this study will receive 2 dose levels of imatinib, 200 mg orally daily followed by 400 mg orally daily.
  Other Names: Gleevec

SUMMARY:
To determine if subjects with steroid refractory cGVHD can tolerate imatinib mesylate and whether their cGVHD responds to imatinib mesylate.

ELIGIBILITY:
INCLUSION CRITERIA

* Chronic graft-vs-host disease (cGVHD) requiring systemic therapy occurring > 100 days after hematopoietic cell transplant with either:

  1. Persistent steroid dependence defined as the inability to taper steroid treatment to less than 0.25 mg/kg/d prednisone or its equivalent for at least 3 months.
  2. Progression of cGVHD signs and symptoms on steroid therapy equivalent to prednisone 0.5 mg/kg/d for at least 1 month.
* At least one of the following manifestations:

  1. Skin changes (rash, sclerosis, fasciitis, or ulceration).
  2. Abnormal eye wetness ≤ 5 mm as measured by Schirmer's test.
  3. Oral mucosal changes (erythema, lichenoid changes, ulcers, or mucoceles).
  4. Thrombocytopenia (platelets < 50,000/uL).
  5. Abnormal liver function testing defined as alkaline phosphatase, AST, ALT, or total bilirubin > upper limit of normal (ULN).
  6. Bronchiolitis obliterans (diagnosed by a > 5% annual decline in FEV1 with the lowest post-transplant FEV1/FVC < 0.8 and an appropriate CT scan or lung biopsy).
* Has been on a fixed dose of steroids or a fixed dose of steroids and one other immunosuppressant (cyclosporine, tacrolimus, sirolimus, mycophenolate mofetil, or extracorporeal photopheresis) for ≥ 30 days before starting imatinib.
* Life expectancy ≥ 6 months.
* Ability to understand and willingness to sign a written informed consent document.
* Karnofsky performance status ≥ 3 50% (Appendix B).
* At least 18 years of age.
* If a female of reproductive potential (defined as having at least 1 menstrual period in the past 12 months), must have a negative pregnancy test performed ≤ 7 days before starting study drug.
* If a female of reproductive potential, agrees to use contraception for the duration of the trial.
* Total bilirubin < 1.5X ULN.
* Aspartate transaminase (AST) < 2.5 x ULN.
* Alanine aminotransferase (ALT) < 2.5 x ULN.
* Alkaline phosphatase < 2.5 x ULN.
* Absolute neutrophil count (ANC) > 500/uL (growth factor supplementation is allowed).
* Hematocrit > 26% (transfusion support is allowed).
* Platelet count > 20,000/uL.

EXCLUSION CRITERIA

* Received another investigational agent ≤ 30 days before starting the study drug.
* Ongoing intercurrent illness such as an infection not responsive to antibiotics, antiviral medicines, or antifungal medicines.
* Progressive malignant disease.
* Secondary malignancy that has not been effectively treated within the past 5 years (except localized basal cell or squamous cell carcinoma).
* Imatinib intolerance or allergy.
* Participant is breast-feeding.
* Not willing to comply with treatment or response evaluation.
* Received an allogeneic cell product [including donor lymphocyte infusion (DLI) or hematopoietic cell boost] ≤ 100 days before starting study drug.
* Steroid and/or immunosuppressant dose has changed ≤ 30 days before starting study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The frequency of adverse events graded according to the CTCAE will be the primary endpoint | Subjects will be monitored at 1, 4, 8, 16, and 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: David Miklos, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - Fred Hutchinson Cancer Research Center (FHCRC), Seattle, Washington

REFERENCES:
- [Result] Chen GL, Arai S, Flowers ME, Otani JM, Qiu J, Cheng EC, McMillan A, Johnston LJ, Shizuru JA, Miklos DB. A phase 1 study of imatinib for corticosteroid-dependent/refractory chronic graft-versus-host disease: response does not correlate with anti-PDGFRA antibodies. Blood. 2011 Oct 13;118(15):4070-8. doi: 10.1182/blood-2011-03-341693. Epub 2011 Aug 9. PMID 21828142